CLINICAL TRIAL: NCT06764693
Title: Prospective Multi-country, Real-world, Multi-arm Study of Treatment PErsistence With RISankizumab in Psoriatic Arthritis (PERIS)
Brief Title: An Ex-US Study to Assess Treatment Persistence With Risankizumab in Adult Participants With Psoriatic Arthritis
Acronym: PERIS
Status: Recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P24-390
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Psoriatic Arthritis
Keywords: Risankizumab, Skyrizi
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Biologic Disease-Modifying Antirheumatic Drugs (bDMARD): Participants will receive bDMARDs as prescribed by their physician according to local label.
- Risankizumab: Participants will receive risankizumab as prescribed by their physician according to local label.

SUMMARY:
Psoriatic arthritis (PsA) is a type of arthritis (swelling and stiffness in the joints) that is frequently seen in trial participants who also have the skin condition psoriasis. It is caused by an overactive immune system where the body attacks healthy tissue by mistake. This study aims to describe the long term usage and effectiveness with risankizumab (RZB) relative to other advanced therapeutic options for the management of PsA in daily clinical practice.

Risankizumab is an approved drug for the treatment of psoriatic arthritis. The study will not be conducted in the United States, however it will be conducted in approximately 15 countries and include at least 900 and up to 1200 participants with a 2 to1 ratio of participant allocation between participants receiving risankizumab and participants receiving other advanced therapeutic agents.

The therapy is prescribed in the usual manner in accordance with the terms of the local marketing authorization and professional and reimbursement guidelines with regards to dose, population, and indication. All study visits will occur during routine clinical practice and participants will be followed for 24 months.

There is expected to be no additional burden for participants in this study.

ELIGIBILITY:
Inclusion Criteria:

* Participant with a clinical diagnosis of psoriatic arthritis (PsA) with symptom onset at least 6 months prior to the Screening visit and fulfillment of ClASsification for Psoriatic ARthritis (CASPAR) at Baseline visit to confirm that the participant has active disease.
* Participant must have demonstrated an inadequate response to at least 1 Disease-modifying antirheumatic drug (DMARD) (with max 50% Biologic DMARD-Inadequate Response); alternatively, participant must have demonstrated an intolerance to or contraindication for csDMARDs as determined by the investigator.

Exclusion Criteria:

- Participants demonstrated an inadequate response to three or more bDMARDs/targeted synthetic DMARDs (tsDMARDs).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants that currently are treated with Risankizumab or other advanced treatment options for the management of active psoriatic arthritis in clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants that show persistence in treatment until 24 months | 24 Months
  Persistence over 24 months, defined as a participant who starts PsA treatment and is still on the same therapy until 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (127):
- Argentina (3):
  - Cer Instituto Médico /ID# 274445, Quilmes, Buenos Aires
  - Instituto Medico de Alta Complejidad San Isidro S.A. /ID# 274417, San Isidro, Buenos Aires
  - Instituto Médico Río Cuarto /ID# 274421, Río Cuarto, Córdoba Province
- Austria (4):
  - Landesklinikum Stockerau /ID# 275618, Stockerau, Lower Austria
  - Medizinische Universitaet Graz /ID# 273765, Graz, Styria
  - Krankenhaus Der Barmherzigen Brueder Graz /ID# 273764, Graz, Styria
  - Rheuma-Zentrum Wien-Oberlaa GmbH /ID# 275617, Vienna, Vienna
- Belgium (7):
  - Universite Libre de Bruxelles - Hopital Erasme /ID# 272763, Anderlecht, Brussels Capital
  - Rhumaconsult Sprl /ID# 272797, Charleroi, Hainaut
  - Reumacentrum Genk - Medisch Centrum Genk /ID# 272796, Genk, Limburg
  - ReumaClinic /ID# 272782, Genk, Limburg
  - OLV Ziekenhuis Aalst /ID# 274456, Aalst, Oost-Vlaanderen
  - UZ Leuven /ID# 272781, Leuven, Vlaams-Brabant
  - CHU de Liege /ID# 272784, Liège
- Bulgaria (6):
  - Diagnostic Consultative Centre (Dcc) - Foкus 5 /ID# 275952, Sofiya, Sofia
  - Military Hospital - Pleven /ID# 276054, Pleven
  - Medical Center Epiona /ID# 276037, Plovdiv
  - Dr. Tsvetanka Petranova ELIMED - 2 /ID# 276158, Sofia
  - Medical Center Academy /ID# 276041, Sofia
  - AIPSMPR -d-r Gerganov /ID# 275953, Varna
- Czechia (2):
  - MAPO revma /ID# 272409, Ostrava, Ostrava-mesto
  - Fakultni Nemocnice Plzen /ID# 276061, Pilsen, Praha 17
- France (27):
  - Centre Hospitalier Universitaire de Nice - Hopital Pasteur /ID# 274923, Nice, Alpes-Maritimes
  - Infirmerie Protestante De Lyon /ID# 274922, Caluire-et-Cuire, Auvergne-Rhône-Alpes
  - Centre Hospitalier Universitaire Gabriel-Montpied /ID# 275399, Clermont-Ferrand, Auvergne-Rhône-Alpes
  - Chu Grenoble - Hôpital Sud /ID# 275200, Échirolles, Auvergne-Rhône-Alpes
  - Centre Hospitalier Régional Universitaire de Besançon - Hôpital Jean Minjoz /ID# 277881, Besançon, Doubs
  - Centre Hospitalier D'Arras /ID# 275192, Arras, Hauts-de-France
  - CHU de Lille - Hôpital Salengro /ID# 274980, Lille, Hauts-de-France
  - Chu Montpellier /ID# 274925, Montpellier, Herault
  - Chru De Rennes - Hôpital Sud /ID# 277115, Rennes, Ille-et-Vilaine
  - Centre Hospitalier Régional Universitaire De Tours - Hôpital Trousseau /ID# 275397, Chambray-lès-Tours, Indre-et-Loire
  - Clinique François Chénieux /ID# 276516, Limoges, Limousin
  - CHU Limoges - Dupuytren 2 /ID# 274918, Limoges, Nouvelle-Aquitaine
  - Pôle Santé du Pont de Chaume /ID# 275608, Montauban, Occitanie
  - Centre Hospitalier Boulogne-Sur-Mer /ID# 277269, Boulogne-sur-Mer, Pas-de-Calais
  - Centre Hospitalier Universitaire de Nantes, Hotel Dieu -HME /ID# 275396, Nantes, Pays de la Loire Region
  - Hôpital Privé De Provence /ID# 275797, Aix-en-Provence, Provence-Alpes-Côte d'Azur Region
  - Centre Hospitalier De Cannes - Hôpital De Cannes /ID# 275193, Cannes, Provence-Alpes-Côte d'Azur Region
  - Centre Hospitalier Universitaire de Rouen (CHU)- Hopital Charles Nicolle /ID# 275366, Rouen, Seine-Maritime
  - Cabinet libéral du Dr PAUPIERE /ID# 275401, Péronne, Somme
  - Henri Mondor Hospital /ID# 275360, Créteil, Val-de-Marne
  - CH de Cahors /ID# 275092, Cahors
  - Centre Hospitalier Régional d'Orléans - Hôpital de la Source /ID# 275377, Orléans
  - AP-HP - Groupe Hospitalier 10e - Hopital Lariboisiere /ID# 275182, Paris
  - Groupe Hospitalier Paris Saint-Joseph /ID# 274981, Paris
  - Centre Hospitalier de Valenciennes /ID# 276354, Valenciennes
  - Centre Hospitalier Sud Francilien /ID# 275038, Corbeil-Essonnes, Île-de-France Region
  - Hopital Pitie Salpetriere /ID# 275368, Paris, Île-de-France Region
- Germany (22):
  - Klinische Forschung Im Medizinischen Versorgungalltag Gbr /ID# 276208, Planegg, Bavaria
  - Private Practice - Dr. Dirk Wernicke /ID# 279748, Hohen Neuendorf, Brandenburg
  - Rheumatologisch Immunologisch /ID# 275832, Templin, Brandenburg
  - Deutsches Endokrinologisches Versorgungszentrum DEVZ - MVZ GdR /ID# 276484, Frankfurt am Main, Hesse
  - Rheumateam Lahn-Dill-Siegerland /ID# 276019, Wetzlar, Hesse
  - Praxis. F. Bigdeli-Wilshusen /ID# 275522, Hanover, Lower Saxony
  - Rheumatologie Kassel /ID# 276311, Kassel, Lower Saxony
  - Rheumazentrum Ratingen /ID# 278190, Ratingen, North Rhine-Westphalia
  - Praxis Dr. med. Florian Beyer /ID# 276233, Kaiserslautern, Rhineland-Palatinate
  - Krankenhaus der Barmherzigen Brüder Trier /ID# 278759, Trier, Rhineland-Palatinate
  - Knappschaftsklinikum Saar /ID# 279850, Püttlingen, Saarland
  - Rheumapraxis Dr. Prothmann /ID# 275712, Püttlingen, Saarland
  - Rheumapraxis Dr. Liebhaber /ID# 276235, Halle, Saxony-Anhalt
  - Rheumatologische Facharztpraxis /ID# 276359, Magdeburg, Saxony-Anhalt
  - Universitaetsklinikum Schleswig-Holstein Campus Luebeck /ID# 275711, Lübeck, Schleswig-Holstein
  - Private Practice - Dr. Jochen Walter /ID# 280067, Rendsburg, Schleswig-Holstein
  - Private Practice - Dr. Thomas Kupka /ID# 276236, Altenburg, Thuringia
  - Rheumapraxis Steglitz /ID# 279413, Berlin
  - Private Practice - Dr. Silke Zinke /ID# 279350, Berlin
  - MVZ Herzogin Elisabeth Hospital /ID# 275583, Braunschweig
  - Praxis Fiene /ID# 279363, Greifswald
  - Cellitinnen-Krankenhaus St. Josef /ID# 275710, Wuppertal
- Greece (16):
  - Olympion General Clinic /ID# 271685, Pátrai, Achaia
  - Athens Naval Hospital /ID# 272313, Athens, Attica
  - General Hospital of Athens Ippokratio /ID# 262528, Athens, Attica
  - General Hospital of Athens Laiko /ID# 272325, Athens, Attica
  - General Hospital of Athens Laiko /ID# 272410, Athens, Attica
  - University General Hospital Attikon /ID# 272358, Athens, Attica
  - Asklipieio General Hospital of Voula /ID# 272326, Voula, Attica
  - University General Hospital of Heraklion /ID# 271743, Heraklion, Crete
  - University General Hospital of Alexandroupolis /ID# 272411, Alexandroupoli, Evros
  - The University Hospital of Larissa /ID# 272315, Larissa, Larisa
  - KAT Atttica General Hospital /ID# 271741, Athens
  - General Hospital of Ioannina G. Hatzikosta /ID# 272327, Ioannina
  - Bioclinic Thessaloniki /ID# 272316, Thessaloniki
  - General Hospital of Thessaloniki Hippokrateio /ID# 272314, Thessaloniki
  - Euromedica General Clinic of Thessaloniki /ID# 272412, Thessaloniki
  - Euromedica General Clinic of Thessaloniki /ID# 275805, Thessaloniki
- Ireland (6):
  - St James Hospital /ID# 260024, Dublin, Dublin
  - St Vincents University Hospital /ID# 261237, Elm Park, Dublin
  - University Hospital Kerry /ID# 266733, Tralee, Kerry
  - Cork University Hospital /ID# 268263, Cork
  - Beaumont Hospital /ID# 271961, Dublin
  - Tallaght University Hospital /ID# 277000, Dublin
- Israel (6):
  - Meir Medical Center /ID# 273315, Kfar Saba, Central District
  - The Chaim Sheba Medical Center /ID# 273313, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 273311, Tel Aviv, Tel Aviv
  - The Lady Davis Carmel Medical Center /ID# 273312, Haifa
  - Hadassah Medical Center-Hebrew University /ID# 273314, Jerusalem
  - Galilee Medical Center /ID# 275431, Nahariya
- Italy (13):
  - IRCCS Istituto Clinico Humanitas /ID# 264463, Rozzano, Lombardy
  - ASST Centro Specialistico Ortopedico Traumatologico Gaetano Pini-CTO /ID# 265161, Milan, Milano
  - IRCCS Ospedale San Raffaele /ID# 266212, Milan, Milano
  - Azienda Ospedaliera Universitaria Luigi Vanvitelli /ID# 266888, Naples, Napoli
  - Azienda Ospedaliero-Universitaria Policlinico Umberto I /ID# 265145, Rome, Roma
  - Azienda Ospedaliero Universitaria delle Marche /ID# 264636, Ancona
  - ASST degli Spedali Civili di Brescia /ID# 264699, Brescia
  - Universita degli Studi del Molise /ID# 265162, Campobasso
  - AOU Policlinico G. Rodolico - San Marco /ID# 264459, Catania
  - ASL 2 Abruzzo Lanciano-Vasto-Chieti /ID# 265640, Chieti
  - Azienda Ospedaliero Universitaria Pisana /ID# 264938, Pisa
  - Azienda Ospedaliera Universitaria Senese /ID# 265207, Siena
  - ASU FC - P.O. Universitario Santa Maria della Misericordia /ID# 264698, Udine
- Poland (2):
  - Indywidualna Specjalistyczna Praktyka Lekarska dr hab.n.med.Katarzyna Pawlak-Buś /ID# 276483, Poznan, Greater Poland Voivodeship
  - SOMED Renata Sokolik /ID# 276480, Wroclaw, Lower Silesian Voivodeship
- Imam Abdulrahman Bin Faisal University /ID# 277716, Dammam, Eastern Province, Saudi Arabia
- Spain (11):
  - Hospital Universitario Virgen de la Victoria /ID# 264317, Málaga, Malaga
  - Hospital Rafael Mendez /ID# 272663, Lorca, Murcia
  - Hospital Xeral Cies (CHUVI) /ID# 272659, Vigo, Pontevedra
  - Hospital Universitario de Valme /ID# 264314, Seville, Sevilla
  - Hospital Universitario Virgen de las Nieves /ID# 275741, Granada
  - Hospital Universitario Clinico San Cecilio /ID# 272665, Granada
  - Hospital Juan Ramón Jiménez /ID# 272667, Huelva
  - Hospital Universitario de La Princesa /ID# 264073, Madrid
  - Hospital Universitario 12 de Octubre /ID# 272660, Madrid
  - Hospital Universitario La Paz /ID# 264316, Madrid
  - Hospital General Universitario Reina Sofía /ID# 272664, Murcia
- Taipei Medical University - Shuang Ho Hospital, Ministry of Health and Welfare /ID# 274352, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P24-390